CLINICAL TRIAL: NCT02123784
Title: Biomarkers for the Surgical Treatment of Rotator Cuff Tears
Acronym: MARK-GEROT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Balgrist University Hospital (Other)
Collaborators: RESORTHO foundation, Forchstrasse 340, 8008 Zürich, Switzerland (Unknown)
Responsible Party: Principal Investigator, Professor Martin Flück, Professor for Muscle Plasticity, Balgrist University Hospital
Other Study IDs: W 522 MARK GEROT; KEK-ZH-Nr. 2013-0352 (Other: Ethics Committee of the Canton Zurich, Switzerland)
Record Dates: First submitted 2014-04-14; First posted 2014-04-28 (Estimated); Last update posted 2016-07-04 (Estimated); Status verified 2016-07

CONDITIONS: Rotator Cuff Tears
Keywords: Rotator Cuff Tear; Rotator Cuff Repair; Biomarker; Predictive factors; Skeletal Muscle; Tendon; Subacromial Bursa
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, muscle, tendon, capsule, synovial liquid
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Rotator cuff tear: Patients which demonstrate a full-thickness tear of the rotator cuff tendon and meet the inclusion criteria.

SUMMARY:
Identification of biomarkers that can predict the outcome of the surgical treatment (i.e. the rate of re-rupture) of tears in the rotator cuff tendon.

DETAILED DESCRIPTION:
Rotator cuff tears (i.e. structural failure and tissue disruption in at least one of the four muscles and tendons that form the rotator cuff) are extremely common injuries and represent the most common muscle-tendon tear in patients. Repair of rotator cuff tears is usually advocated for painful tears with functional impairment. However, high failure rates of 13-68% have been reported for surgical repair of rotator cuff tears, irrespective of the surgical technique employed. Higher rates of re-rupture are associated with larger tears, increased patient age, and increased fatty degeneration of the cuff muscles. There is no general consensus as to the causes of re-rupture; where mechanical factors, the existing techniques of suturing, and biological factors are considered as the main factors of recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Full-thickness rotator cuff tear (isolated transmural supraspinatus muscle tear or combined with infraspinatus and subscapularis tears) with fat content <50% (Goutallier stage 0-2), as confirmed by magnetic resonance imaging
* Acute or chronic ruptures
* Older than 40 years of age
* Voluntary participation in this study
* Written informed consent to participate in this study

Exclusion Criteria:

* Contraindication because of ethical reasons
* Pregnant or lactating women
* Intention/wish to become pregnant during the course of this study
* Unsafe contraception
* Clinical co-morbidities, such as renal insufficiency, hepatic dysfunction, cardiovascular disease
* Known or suspected non-adherence to the study protocol
* Smoker
* Drug or alcohol addicted
* Uncapable of following instructions, e.g. because of insufficient proficiency in languages, psychological problems, dementia, etc.
* Participation in other clinical trials during the duration of this study, as well as 30 d before inclusion in this study
* Claustrophobia
* Systemic corticoid steroid therapy

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Regular patients from Balgrist University Hospital, Zurich (Switzerland)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-04; Primary Completion 2017-06 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline for anatomical and functional characteristics of the ruptured rotator cuff | Before surgery (baseline), 3 months after surgery, 12 months after surgery
  Patients will undergo a clinical and functional examination which includes the assessment of mobility, pain and abduction force of the affected and healthy shoulder using standardized tests (Constant score, Quick DASH, Quality of Life Score SF-12), the quantification of the volume (cm3) and fat content (Goutallier Stage) of the affected shoulder using magnet resonance imaging.
Molecular and cellular characteristics of the tissues affected by tears of the rotator cuff | within 1 year after the last surgery
  Before the surgery 10 mL of venous blood will be drawn from the patients and processed for the isolation of genomic DNA and the measure of selected single nuclear polymorphisms.
  Biopsies (~10 mg) will be collected intra-operatively from the affected muscle, tendon, capsule and synovial liquid and stored at -80°C. Samples will be subjected to the immunohistochemical and biochemical quantification of the content (in arbitrary units) of selected proteins and tissue composition (as % of total volume).

SECONDARY OUTCOMES:
Correlation between the molecular and cellular characteristics at the point in time of surgery, and the clinical (magnetic resonance imaging) outcomes | within 1 year after the last surgery
  The relationship of the molecular and cellular parameters (measured as primary endpoints) of affected muscle with the clinical and functional measures of shoulder function will be investigated using Pearson correlation and mutual information analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Balgrist University Hospital, Zurich, Switzerland

REFERENCES:
- [Derived] Olthof MGL, Fluck M, Borbas P, Valdivieso P, Toigo M, Egli F, Joshy J, Filli L, Snedeker JG, Gerber C, Wieser K. Structural Musculotendinous Parameters That Predict Failed Tendon Healing After Rotator Cuff Repair. Orthop J Sports Med. 2023 Sep 19;11(9):23259671231196875. doi: 10.1177/23259671231196875. eCollection 2023 Sep. PMID 37736603